CLINICAL TRIAL: NCT01423838
Title: Comparison of Oxybutynin and Solifenacin in the Treatment of Overactive Bladder: a Randomized Controlled Multicenter Trial
Brief Title: Comparison of Solifenacin and Oxybutynin in the Treatment of Overactive Bladder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adana Numune Training and Research Hospital (Other Government)
Collaborators: Kocaeli University (Other); Akdeniz University (Other); Cukurova University (Other); Baskent University (Other); Ankara University (Other); University of Gaziantep (Other); Inonu University (Other); Gaziosmanpasa University (Unknown); Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Murat Api, Associate Professor, M.D., Ph.D., Adana Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Solifenacin vs Oxybutynin
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; Solifenacin; Oxybutynin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Solifenacin (Active Comparator): Anticholinergic molecule used in the treatment of overactive bladder.
  Interventions: Drug: Solifenacin
- Oxybutynin (Active Comparator): Anticholinergic molecule used in the treatment of overactive bladder.
  Interventions: Drug: Oxybutynin

INTERVENTIONS:
Drug: Solifenacin — 5 mg, oral, once in a day
  Other Names: Kinzy
  Arms: Solifenacin
Drug: Oxybutynin — 5 mg, oral, three times in a day
  Other Names: Uropan
  Arms: Oxybutynin

SUMMARY:
Null hypothesis of the trial is that there is no difference between solifenacin and oxybutynin with respect to efficacy, side effects, patient satisfaction and quality of life measures in patients with overactive bladder.

DETAILED DESCRIPTION:
In this two-month follow-up study, the patients with overactive bladder will be randomly assigned into two groups (solifenacin or oxybutynin in their usual doses) and will be assessed with respect to baseline characteristics and complaints before treatment. After initiation of the treatment at first and second months follow-up visits the patients will be reassessed with respect to compliance, satisfaction, degree of improvement, reasons for dropouts, number and severity of side effects.

ELIGIBILITY:
Inclusion Criteria: Women between 18-70 years of age, diagnosed to have overactive bladder (presence of at least two of the following three main criteria: urgency, urge incontinence, frequency and nocturia)

Exclusion Criteria: Presence of stress urinary incontinence, patients who are still using a drug for overactive bladder, pregnant women, women in postpartum period (women on lactation), patients who have closed angle glaucoma, patients with chronic constipation, having allergy to the ingredients of the drugs, patients having the contraindicated conditions listed in the printed instructions of the drugs.

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement in overactive bladder symptoms | 2 months
  The main symptoms of overactive bladder are frequency, urgency, urge incontinence and nocturia (if any). The primary outcome of the trial will be comparison of the improvement of these symptoms in terms of number and severity between two study groups.

SECONDARY OUTCOMES:
To compare the degree of side effects between two study groups | 2 months
  Outcome measures will be compliance to the study drugs, patient satisfaction, willingness to continue treatment, degree of side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Api, M.D., Ph.D., Study Director — Turkish Republic Ministry of Health Adana Numune Training and Research Hospital
Locations (1):
- Turkish Republic Ministry of Health Adana Numune Training and Research Hospital, Adana, Turkey (Türkiye)